CLINICAL TRIAL: NCT01935713
Title: Novel Methods to Reduce Children's Secondhand Smoke Exposure I
Brief Title: Preliminary Investigation of Novel Methods to Reduce Children's Secondhand Smoke Exposure
Acronym: EZI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EZ Study
Record Dates: First submitted 2013-08-30; First posted 2013-09-05 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Secondhand Smoke
MeSH Terms: interventions — Tobacco Use Cessation Devices; Nicotine Chewing Gum; Electronic Nicotine Delivery Systems

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Electronic Cigarette (Experimental): Participants received the electronic cigarette for use instead of cigarettes when in the presence of their child(ren) for up to 8 weeks.
  Interventions: Drug: Electronic Cigarette
- Dissolvable Tobacco Lozenge (Experimental): Participants received the dissolvable tobacco lozenge for use instead of cigarettes when in the presence of their child(ren) for up to 8 weeks.
  Interventions: Drug: Dissolvable Tobacco Lozenge
- Dissolvable Nicotine Lozenge (Nicorette) (Experimental): Participants received the dissolvable nicotine lozenge (Nicorette) for use instead of cigarettes when in the presence of their child(ren) for up to 8 weeks.
  Interventions: Drug: Nicotine polacrilex

INTERVENTIONS:
Drug: Nicotine polacrilex — Participants were given the choice of 2mg or 4mg lozenges depending on how many cigarettes per day they reported to smoke.
  Other Names: Nicorette
  Arms: Dissolvable Nicotine Lozenge (Nicorette)
Drug: Electronic Cigarette — Participants were given an e-cigarette starter kit, charging case, and cartridges in either 12mg or 16 mg nicotine, depending on their current amount of cigarettes smoked per day.
  Other Names: Smoke Tip
  Arms: Electronic Cigarette
Drug: Dissolvable Tobacco Lozenge — Participants were given Ariva (light to moderate smokers) or Stonewall (heavier smokers, >2 packs per day).
  Other Names: Ariva, Stonewall
  Arms: Dissolvable Tobacco Lozenge

SUMMARY:
The overall aim of the current study is to determine if the use of nicotine containing products by caregivers who smoke and who are not interested in quitting, is effective in reducing children's secondhand smoke exposure.

ELIGIBILITY:
Inclusion Criteria: In order to be included in the study, participants must:

1. be the primary caregiver(defined as a person who spends the most time with the child and spends a minimum of 4 hours per day in the presence of the child) of a child between the ages of 3-11 (if caregiver has more > 1 child between 3-11 years, we will include the youngest)
2. smoke at least 10 cigarettes per day for the past year
3. indicate that they smoke around their child or in the car or home at least one time per week]
4. have no intention of quitting smoking in the next 12-weeks
5. aged 18-65 years
6. be fluent in English
7. have no recent history of cardiovascular distress that may contraindicate medicinal nicotine lozenge use (heart attack in the past year, arrhythmia, uncontrolled hypertension)
8. not currently pregnant, planning to become pregnant, or breastfeeding
9. do not use non-cigarette tobacco (cigars, chewing tobacco)
10. have no prior use of any potential reduced exposure product
11. have no major psychiatric impairment, including psychosis, suicidality, and/or any current alcohol/drug abuse or dependence

Exclusion Criteria:

* Does not meet all of the requirements of inclusion criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2012-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in child salivary cotinine | 2, 4, 8, and 12 weeks
  Child salivary cotinine will be measured to assess the level of secondhand smoke exposure. We will measure the change throughout the study.

SECONDARY OUTCOMES:
Change in Parent and Child Lung Function | 2, 4, 8, and 12 weeks
  We will collect both parent and child spirometry data and compare changes.

CONTACTS AND LOCATIONS:
Locations (1):
- The Children's Hospital at OU Medical Center, Oklahoma City, Oklahoma, United States